CLINICAL TRIAL: NCT01039532
Title: Comparison of Thrice Daily Biphasic Human Insulin Versus Basal Detemir and Bolus Aspart in Patients With Poorly Controlled Type 2 Diabetes Mellitus
Brief Title: Comparison of Thrice Daily Biphasic Human Insulin With Basal Bolus Regimen in Type 2 Diabetes Mellitus Patients
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Anil Bhansali, prof and head, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Other Study IDs: BHI3
Record Dates: First submitted 2009-12-24; First posted 2009-12-25 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes mellitus; Biphasic human insulin thrice a day; Basal bolus insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Basal Bolus regimen: Basal Bolus regimen
- Biphasic human insulin: Biphasic human insulin

SUMMARY:
It is a proven fact that Basal Bolus insulin regimen is the near- physiological regimen & Thrice daily Biphasic Insulin Aspart is a comparable alternative for glycemic control in type 2 diabetes mellitus patients. In this study the investigators evaluated whether Biphasic Human Insulin can be used in a thrice daily regimen in place of BIAsp.

As the regimen is less expensive and one prick less than the basal-bolus regimen, it can be a good alternative for a diabetics in India.

This is a 12 week Open labelled parallel-Randomised controlled pilot study - 50 patients with type 2 Diabetes mellitus was selected after satisfying the inclusion and exclusion criteria's .Metformin and pioglitazone were continued and they are randomised into 2 groups at base line and was allotted into any of the two regimens.

1. Basal detemir + bolus aspart or
2. Thrice Daily Biphasic Human Insulin Regimen.

The two regimens were compared by the following variables:

Primary endpoint:

Glycaemic control

Secondary endpoint:

Weight gain, Hypoglycaemic episodes, Adverse effects and Cost effectiveness

DETAILED DESCRIPTION:
It is a proven fact that Basal Bolus insulin regimen is the near- physiological regimen & Thrice daily Biphasic Insulin Aspart is a comparable alternative for glycemic control in type 2 diabetes mellitus patients. In this study the investigators evaluated whether Biphasic Human Insulin can be used in a thrice daily regimen in place of BIAsp.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetics >/= 18 yrs of age Diabetic for >/= 6months
* Inadequately controlled patients treated with human premixed insulin twice daily for at least 3months along with metformin 2g/d and pio30mg/d

  * Single dose of insulin exceeding 25 units or total insulin dose is more than 0.7u/kg/day with
  * If post lunch blood glucose is not controlled
  * If HbA1c ≥7%
* No major cardiac events in the preceding 6 months.
* NYHA <= Class II.

Exclusion Criteria:

* Deranged LFT's- AST,ALT or ALP values >= 2 times.
* Deranged RFT Sr. Creatinine >=1.5
* Allergy to Insulin or its products.
* Recent intake of any new medications for sugar control.
* Illiterate to the level that she/he cannot understand the study.
* Any other acute co morbid illness.
* Pregnancy.
* Decompensated heart failure/UsA/MI all within last 12month
* Untreated proliferative retinopathy/ maculopathy
* Drug or alcohol dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 type 2 diabetes mellitus patients inadequately controlled patients treated with human premixed insulin twice daily for at least 3months along with metformin 2g/d and pioglitazone 30mg/d.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Glycaemic control | 3months

SECONDARY OUTCOMES:
Weight gain Hypoglycaemic episodes Adverse effects Cost effectiveness | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anil Bhansali, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- AnilBhansali, Chandigarh, Chandigarh, India